CLINICAL TRIAL: NCT05648799
Title: Multicenter Open Two-stage Study of Pharmacokinetics, Safety and Efficacy of GP30341, 200 mg Capsules (GEROPHARM LLC, Russia) in Healthy Volunteers and Outpatients With Novel Coronavirus Infection 2019 With a High Risk of Adverse Outcome
Brief Title: Pharmacokinetics, Safety and Efficacy Study of GP30341 (GEROPHARM, Russia)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP30341-P4-31
Record Dates: First submitted 2022-12-07; First posted 2022-12-13 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2022-10

CONDITIONS: Pharmacokinetics; Safety Issues; Efficacy
Keywords: Molnupiravir; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir; Standard of Care

STUDY DESIGN:
Intervention Model Description: two-stage study: 1 stage - two-period escalating dose study involved two sequential cohorts of 6 healthy volunteers. 2 stage - randomized comparative study with hypothesis of superior efficacy in parallel groups.
Masking Description: This study was conducted as open to the Participant and the Investigator. However, collected blood samples were blinded to an analytical laboratory specialist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP30341 capsules 200 mg (Experimental): 4 capsules containing 200 mg of molnupiravir p.o. twice a day during 5 days (daily dose 1600 mg) in combination with Standard therapy in accordance with the current version of the guidelines for the prevention, diagnosis and treatment of a new coronavirus infection 2019 (COVID-19).
  Interventions: Drug: GP30341 capsules 200 mg
- Standart therapy (Active Comparator): Standard therapy in accordance with the current version of the guidelines for the prevention, diagnosis and treatment of a new coronavirus infection 2019 (COVID-19).
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: GP30341 capsules 200 mg — orall take of capsules twice a day
  Other Names: molnupiravir
  Arms: GP30341 capsules 200 mg
Drug: Standard therapy — Standard medicines for treatment of a new coronavirus infection 2019 (COVID-19).
  Other Names: COVID-19 therapy
  Arms: Standart therapy

SUMMARY:
Pharmacokinetics, safety and efficacy study of GP30341, 200 mg capsules (GEROPHARM LLC, Russia) in healthy volunteers and patients with novel coronavirus infection 2019 (COVID-19) with a high risk of adverse outcome

DETAILED DESCRIPTION:
Multicenter open two-stage study of pharmacokinetics, safety and efficacy of GP30341, 200 mg capsules (GEROPHARM LLC, Russia) involving healthy volunteers and patients with novel coronavirus infection 2019 (COVID-19) with a high risk of adverse outcome.

I stage: An open non-comparative study of pharmacokinetics and safety of GP30341 studied at different dosing regimens with an escalation of the daily dose in healthy volunteers.

II stage: Open randomized study efficacy and safety of GP30341, 200 mg capsules with active control - comparison with standard therapy - in patients with COVID-19 infection with a high risk of adverse outcome.

ELIGIBILITY:
Stage 1

Inclusion Criteria:

* Signed informed consent to participate in the study.
* Males with a verified diagnosis "healthy" according to the data of standard clinical, laboratory and instrumental examination methods.
* Age 18-45 years old inclusive.
* Body mass index 18.5 - 30 kg/m2.
* Agree to use an adequate method of contraception (double barrier method) during the entire period of participation in the study and for 3 weeks after its completion.
* Consent to all restrictions imposed during the study.
* Citizenship of the Russian Federation.

Exclusion Criteria:

* Burdened allergic history, drug intolerance.
* Hypersensitivity to heparin, molnupiravir and any of the excipients of the study drug.
* Any acute and chronic diseases, incl. but not limited to:

  1. diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract (including diseases of the colon), liver, kidneys, blood;
  2. positive test results for hepatitis C (antibodies) or hepatitis B (surface antigen), HIV (antibodies to HIV-1/2), syphilis (antibodies to Treponema pallidum).
* Deviations from normal values of heart rate (60-89), SBP (90-130 mm Hg), DBP (60-89 mm Hg), NPV (12-20), body temperature (35.7 - 37.0 °C).
* ECG Deviations, according to a specialist, during screening.
* laboratory tests results deviations from the normal values.
* Hard-to-reach veins of the upper extremities, vein thrombosis, thrombophlebitis in a family history of close relatives, "compromised" veins due to frequent previous venipunctures.
* Surgical interventions on the gastrointestinal tract (with the exception of appendectomy) in history.
* Acute infectious diseases less than 4 weeks prior to screening.
* Presence of at least one of the epidemic signs:

  1. return from overseas travel 14 days prior to screening and no test results for SARS-CoV-2 RNA or SARS-CoV-2 antigen;
  2. close contact in the last 14 days prior to screening with a person under observation for COVID-19 who subsequently fell ill;
  3. close contact in the past 14 days prior to screening with individuals who have laboratory-confirmed case of COVID-19;
  4. Occupational contacts in the past 14 days prior to screening with individuals who have a suspected or confirmed case of COVID-I9.
* Regular intake of any medications, including vitamins, herbal preparations, and dietary supplements, less than 2 weeks before screening.
* Significant blood loss (more than 450 ml of blood or plasma) within 3 months prior to screening, due to, including, but not limited to, blood donation, blood loss during advanced surgery or trauma.
* Drinking alcohol in quantities exceeding 10 units per week (on average) (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of dry wine or 50 ml of strong alcoholic drinks) or anamnestic information about alcoholism, drug addiction, abuse of strong drugs.
* Positive test results for alcohol, drug use and the use of strong drugs.
* Nicotine addiction (regular tobacco use, including smoking of all types of electronic cigarettes, hookahs, snuff, etc. less than 6 months prior to screening).
* Participation in a clinical trial of any drugs (including experimental drugs) or experimental medical devices for 3 months or 5 half-lives prior to Screening, whichever is longer.
* Dehydration due to diarrhea, vomiting, or other cause within the last 24 hours prior to screening.
* Any diet (eg vegetarian, fasting, etc.) or lifestyle (including night work and extreme physical activity such as heavy lifting) that may interfere with the study.
* Taking drugs that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 30 days before screening.
* Mental diseases, history of epilepsy, seizures.
* Volunteers who are obviously or likely, in the opinion of the investigator, unable to understand and evaluate the information on this study as part of the informed consent process, in particular regarding expected risks and possible discomfort.

Stage2:

Inclusion Criteria:

* Signed informed consent to participate in the study.
* Male and female patients aged ≥18 years at the time of providing informed consent.
* Laboratory confirmation of COVID-19 infection ≤5 days prior to randomization1, defined as a positive RT-PCR test for SARS-CoV-2 RNA and/or a positive antigen test for SARS-CoV-2 in a nasal swab.
* Clinical onset of COVID-19 infection (as ≥1 symptom consistent with COVID-19) ≤5 days prior to randomization.
* Presence of ≥1 symptom consistent with COVID-19 at time of randomization3.
* Mild to moderate COVID-19 infection with ≥1 risk factor for adverse outcome.
* WHO (World Health Organization) Clinical Progression Scale score ≥3 at screening 6.
* Consent and ability to take oral medications.
* Agree to use reliable contraceptive measures throughout the study and for 3 weeks after - Negative pregnancy test in women capable of childbearing.
* Consent and ability to comply with the Protocol's procedures, prohibitions and restrictions.

Exclusion Criteria:

* Hypersensitivity or intolerance reactions to any of the components of the test drug or the proposed standard therapy drugs according to the anamnesis.
* Vaccination to prevent COVID-19 within 6 months prior to screening or planning vaccination during the study period.
* Vaccination with any vaccine within 4 weeks prior to screening.
* Use of drugs from the list of prohibited therapy (section 5.3.3 of the Study Protocol) in the anamnesis or their planned use during the study period.
* Past infection with COVID-19 within 6 months prior to screening.
* Current hospitalization or, in the opinion of the Investigator, expected hospitalization within 48 hours after randomization.
* Dysfunction of organs that affect the absorption and metabolism of the test drug, which include, but are not limited to the following:

  1. diseases of the gastrointestinal tract, which, in the opinion of the researcher, may interfere with the absorption of the contents of the capsules;
  2. Kidney Disease Outcomes Quality Initiative (KDOQI) stage 4 or 5 chronic kidney disease;
* Signs of significant uncontrolled comorbidity, such as disorders of the nervous, respiratory, cardiovascular, kidney, liver, endocrine, or gastrointestinal tract, that persist at the time of screening and, in the opinion of the Investigator, significantly increase the risk of adverse outcome and preclude participation patient in the study.
* Acute pancreatitis or exacerbation of chronic pancreatitis ≤3 months prior to randomization.
* Severe immunodeficiency states, which include, but are not limited to, the following:

  1. HIV infection, syphilis;
  2. chemotherapy within 5 weeks prior to screening;
  3. absolute number of neutrophils in blood <500/mm3;
  4. history of hematopoietic stem cell transplantation.
* Signs of severe or extremely severe COVID-19 infection at the time of screening and randomization.
* Heart rate less than 50 beats per minute at rest at screening.
* Platelet count <100,000/µl or platelet transfusion within 5 days prior to randomization12.
* Pregnancy or lactation in women.
* Alcoholism or alcohol consumption in excess of:

  1. for men: 14 units per week (on average);
  2. for women: 7 units per week (on average).
* Addiction and/or substance abuse.
* Participation in other clinical trials within 28 days prior to screening, or planned participation during the period of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
AUC0-t | cohort N1 -10 minutes, 10, 20, 30, 45 mintes, 1 hour, 1hour 15 minutes, 1.5, 2, 2.5, 4, 5, 6, 8, 10, 12, 24 hours; Cohort N2 -10 minutes, 30 minutes, 1 hour, 2, 12, 12.5, 13, 14, 24, 36 hours
  Total area under the curve "concentration of the active metabolite of the active substance - time" in the time interval from 0 (the moment of taking the drug) to the collection of the last blood sample with the determined concentration of the active substance at the time point t.
Cmax | cohort N1 - 10 minutes, 10, 20, 30, 45 minutes, 1hour, 1hour 15 minutes, 1.5 hour, 2, 2.5, 4, 5, 6, 8, 10, 12, 24 hours; Cohort N2 -10 minutes, 30 minutes, 1hour, 2, 12, 12.5, 13, 14, 24, 36 hours
  maximum concentration of the active metabolite of the active substance in the blood plasma of volunteers during the observation period.
tmax | cohort N1 -10 minutes, 10, 20, 30, 45 minutes, 1hour, 1hour 15 minutes, 1.5hour, 2, 2.5, 4, 5, 6, 8, 10, 12, 24 hours; Cohort N2 -10 minutes, 30 minutes, 1hour, 2, 12, 12.5, 13, 14, 24, 36 hours
  time to reach the maximum concentration (Cmax) of the active metabolite of the active substance in the blood plasma of volunteers.
t1/2 | 0-24 hours
  half-life of the active metabolite of the active substance.
λz | cohort N1 -10 minutes, 10, 20, 30, 45 mintes, 1 hour, 1hour 15 minutes, 1.5, 2, 2.5, 4, 5, 6, 8, 10, 12, 24 hours; Cohort N2 -10 minutes, 30 minutes, 1 hour, 2, 12, 12.5, 13, 14, 24, 36 hours
  rate constant of elimination of the active metabolite of the active substance.
AUC0-∞ | cohort N1 -10 minutes, 10, 20, 30, 45 mintes, 1 hour, 1hour 15 minutes, 1.5, 2, 2.5, 4, 5, 6, 8, 10, 12, 24 hours; Cohort N2 -10 minutes, 30 minutes, 1 hour, 2, 12, 12.5, 13, 14, 24, 36 hours
  total area under the curve "concentration of the active metabolite of the active substance - time" in the time interval from 0 (the moment of taking the drug) to infinity.
Frequency of COVID-19 progression on Day 14 | day 14 from randomization
  Frequency of COVID-19 progression to a more severe severity compared to baseline on Day 14

SECONDARY OUTCOMES:
Proportion of patients hospitalized or dying within 28±2 days of randomization. | 0-30 days from randomization
  Proportion of patients hospitalized or dying from any cause within 28±2 days of randomization.
Proportion of patients with a score of more than 3 on the WHO Clinical Progression Scale on Day of end of therapy, Day 10 and Day 14. | 0-14 days from randomization
  Proportion of patients with a score of more than 3 on the WHO (World Health Organization) Clinical Progression Scale on Day of end of therapy, Day 10 and Day 14.
Time to clinical improvement in the form of a persistent reduction in the number of symptoms characteristic of COVID-19 infection by one or more within 28 ± 2 days from randomization. | 0-30 days from randomization
  Time to clinical improvement in the form of a persistent reduction in the number of symptoms characteristic of COVID-19 infection by one or more within 28 ± 2 days from randomization.
Time to clinical progression in the form of (whichever is sooner) a persistent increase in the number of symptoms characteristic of COVID-19 infection by one or more, hospitalization or death from any cause within 28±2 days from randomization. | 0-30 days from randomization
  Time to clinical progression in the form of (whichever is sooner) a persistent increase in the number of symptoms characteristic of COVID-19 infection by one or more, hospitalization or death from any cause within 28±2 days from randomization.
Proportion of patients with a positive nasal swab test for SARS-CoV-2 on Days 3, Day of end of therapy, 10, 14, 28±2 from randomization. | 0-30 days from randomization
  roportion of patients with a positive nasal swab test for SARS-CoV-2 on Days 3, Day of end of therapy, 10, 14, 28±2 from randomization.

OTHER OUTCOMES:
Percentage of volunteers with AEs associated with the test drug. | 0-30 days from randomization
  Percentage of volunteers with AEs associated with the test drug.
Proportion of CTCAE Grade 5.0 or greater adverse events associated with the test product. | 0-30 days from randomization
  Proportion of CTCAE Grade 5.0 or greater adverse events associated with the test product (probable or definite causation, according to the Principal Investigator).
Proportion of cases of early termination of participation in the study due to the development of adverse events. | 0-30 days from randomization
  Proportion of cases of early termination of participation in the study due to the development of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Noskov, MD, Pr., Principal Investigator — Yaroslavl State Institution of Healthcare "Clinical Hospital No. 3" II stage; Elizaveta Antonova, Principal Investigator — St. Petersburg State Institution of Health Care "City Polyclinic No. 112"; Vladimir Rafalsky, MD, Pr., Principal Investigator — Clinical Research Center of Kaliningrad State Healthcare Institution "Central City Clinical Hospital"; Lubov Shpagina, MD, Principal Investigator — Novosibirsk State Medical University, Ministry of Health of the Russian Federation; Viktor Filimonov, MD, Pr., Principal Investigator — Ryazan State Medical University Ministry of Health of the Russian Federation
Locations (5):
- Russia (5):
  - Kaliningrad State Healthcare Institution "Central City Clinical Hospital", Kaliningrad
  - Novosibirsk Federal State Medical University, Novosibirsk
  - Federal Ryazan State Medical University named after Academician I.P. Pavlov, Ryazan
  - St. Petersburg State Health Institution "City Polyclinic No. 112", Saint Petersburg
  - Yaroslavl Region "Clinical Hospital No. 3", ,, Mayakovskogo st., 61, Yaroslavl

IPD SHARING:
Plan to Share IPD: No